CLINICAL TRIAL: NCT05483660
Title: A Randomized, Controlled, Double-blind Trial on the Efficacy of Gastric Probiotics in the Treatment of Helicobacter Pylori Infection
Brief Title: A Clinical Trial on the Efficacy of Gastric Probiotics in the Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2022-252
Record Dates: First submitted 2022-07-24; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Gastric Probiotics; Side-effect; Eradication rate; Helicobacter pylori
MeSH Terms: interventions — exopolysaccharide biopolymer, Bacillus coagulans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The person in charge of assigning patients to treatment groups does not know which treatments the patients receive, so they do not select patients in order of their own volition.
  Patients themselves do not know what treatment they are receiving, so they do not change their compliance or reporting of symptoms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lactobacillus plantarum (Experimental): 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Interventions: Other: Lactobacillus plantarum
- Bacillus coagulans (Experimental): 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Interventions: Other: Bacillus coagulans
- Lactobacillus plantarum + Bacillus coagulans (Experimental): 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Interventions: Other: Lactobacillus plantarum + Bacillus coagulans
- Placebo (Placebo Comparator): Adult milk powder 15 g per time, three times daily and half an hour before meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lactobacillus plantarum — 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Arms: Lactobacillus plantarum
Other: Bacillus coagulans — 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Arms: Bacillus coagulans
Other: Lactobacillus plantarum + Bacillus coagulans — 1.5×10^10 CFU probiotics and adult milk powder 15g per time , three times daily and half an hour before meal.
  Arms: Lactobacillus plantarum + Bacillus coagulans
Other: Placebo — Adult milk powder 15 g pertime, three times daily and half an hour before meal.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Lactobacillus plantarum, Bacillus coagulans and Lactobacillus plantarum + Bacillus coagulans for eradication of Helicobacter Pylori, as well as the efficacy of Lactobacillus plantarum and Bacillus coagulans on side-effect caused by Helicobacter Pylori.

DETAILED DESCRIPTION:
All patients included in this randomized controlled clinical trial will be selected according to strict inclusion and exclusion criteria. At the same time, the benefits and risks of participating in this trial will be explained to the patients before the start of the study, the patients' right to informed consent will be respected, and the informed consent will be signed. After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner (participants and investigator) in a 1:1:1:1 ratio to Lactobacillus plantarum (1.5×10^10 per time, three times daily) or Bacillus coagulans (1.5×10^10 per time, three times daily) or Lactobacillus plantarum + Bacillus coagulans (1.5×10^10 per time, three times daily) or placebo ( 15g per time, three times daily). At the same time, volunteers will be recruited from healthy people to perform the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* Diagnosed by 13C-UBT within 2 weeks before entry.

Exclusion Criteria:

* Previous treatment for H. pylori infection.
* Administration of antibiotics, probiotics/prebiotics, PPIs, H2 receptor antagonists, bismuth preparations, laxatives, anti-diarrhoeals, and certain antimicrobial traditional Chinese medicines 4 weeks before.
* Previous history of gastrointestinal surgery.
* Severe or unstable diseases.
* Pregnancy or lactation.
* Alcoholics and drug abusers.
* Staff of this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori | The eighth week of the trial
  All participants will have a 13C-urea breath test to see if their 13C value falls below the threshold for H. pylori eradication.

SECONDARY OUTCOMES:
The condition of gastrointestinal symptoms before the trial | Baseline
  We will use Gastrointestinal symptoms rating scale (GSRS) to know about the baseline level of their gastrointestinal symptoms before they receive the probiotic or placebo.
The condition of gastrointestinal symptoms in the first week | The first week of the trial.
  We will use Gastrointestinal symptoms rating scale (GSRS) to know about the level of their gastrointestinal symptoms after they receive the probiotic or placebo already a week.
The condition of gastrointestinal symptoms in the second week | The second week of the trial.
  We will use Gastrointestinal symptoms rating scale (GSRS) to know about the level of their gastrointestinal symptoms after they receive the probiotic or placebo after two weeks.
The condition of gastrointestinal symptoms in the third week | The third week of the trial.
  We will use Gastrointestinal symptoms rating scale (GSRS) to know about the level of their gastrointestinal symptoms after they receive the probiotic or placebo after three weeks.
The condition of gastrointestinal symptoms in the fourth week | The fourth week of the trial.
  We will use Gastrointestinal symptoms rating scale (GSRS) to know about the level of their gastrointestinal symptoms at the fourth week of this trial.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after August 31, 2025, and will be permanently public.
Access Criteria: Everyone